CLINICAL TRIAL: NCT00493415
Title: The Evaluation of the Effect of Nitroglycerine Versus Placebo on the Microcirculation by Means of SDF Imaging in Septic Patients on the ICU
Brief Title: The Effect of Nitroglycerine on Microcirculatory Abnormalities During Sepsis
Acronym: NISMIS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Frisius Medisch Centrum (Other)
Responsible Party: EC Boerma, Medical Center Leeuwarden
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TPO 436; ABR 12558; Eudract 2006-004298-88; CCMO NL12558.099.06
Record Dates: First submitted 2007-06-27; First posted 2007-06-28 (Estimated); Last update posted 2008-07-16 (Estimated); Status verified 2008-07

CONDITIONS: Sepsis; Septic Shock
Keywords: microcirculation; sepsis; nitroglycerine; SDF imaging
MeSH Terms: conditions — Sepsis; Shock, Septic | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): nitroglycerine iv
  Interventions: Drug: nitroglycerin iv
- 2 (Placebo Comparator): nacl 0.9% 4 ml/h iv in the first 30 minutes, 2 ml/h iv in the next 23 hours and 30 minutes
  Interventions: Drug: placebo = nacl 0.9%

INTERVENTIONS:
Drug: nitroglycerin iv — loading dose of 4mg/h iv in the first 30 minutes, 2 mg/h iv in the next 23 hours and 30 minutes
  Other Names: nitropohl
  Arms: 1
Drug: placebo = nacl 0.9% — 4 ml/h iv in the first 30 minutes, 2 ml /h iv in the next 23 hours and 30 minutes
  Other Names: isotonic saline
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the effect of nitro-glycerine on the microcirculation (smallest vessel type) in patients with severe sepsis and septic shock.

Nitro-glycerine is a well known medicine in cardiology and is used to improve circulation. In this ICU the investigators use nitro-glycerine to improve the organ perfusion; but it's no common therapy in the rest of the world. The investigators now compare nitro-glycerine and placebo by looking to the sublingual microcirculation by a small camera (SDF imaging).

DETAILED DESCRIPTION:
This study starts at admission of the patient on the ICU. In the next 24 hours the patient receives nitro-glycerine or placebo (randomised). At time = 0, ½, 2, 12 and 24 hour we evaluate the microcirculation by SDF imaging and monitoring of hemodynamic parameters.

Informed consent is obtained of the relatives.

ELIGIBILITY:
Inclusion Criteria:

* Severe sepsis
* Proven infection
* Informed consent

Exclusion Criteria:

* Age < 18 years
* Pregnancy
* Use of nitroglycerine within 24 hours prior to ICU admittance
* Necessity to use nitroglycerine iv for instable angina

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2007-06; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
increase of MFI by nitro-glycerine | 2 years

SECONDARY OUTCOMES:
decrease of length of stay decrease of SOFA decrease of morbidity/mortality | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: E C Boerma, MD, Principal Investigator — Frisius Medisch Centrum
Locations (1):
- Medical Centre Leeuwarden - Intensive Care Unit, Leeuwarden, Netherlands

REFERENCES:
- [Derived] Boerma EC, Koopmans M, Konijn A, Kaiferova K, Bakker AJ, van Roon EN, Buter H, Bruins N, Egbers PH, Gerritsen RT, Koetsier PM, Kingma WP, Kuiper MA, Ince C. Effects of nitroglycerin on sublingual microcirculatory blood flow in patients with severe sepsis/septic shock after a strict resuscitation protocol: a double-blind randomized placebo controlled trial. Crit Care Med. 2010 Jan;38(1):93-100. doi: 10.1097/CCM.0b013e3181b02fc1. PMID 19730258